CLINICAL TRIAL: NCT01043757
Title: A Randomized Controlled Trial of Financial Incentives for Increasing Exercise
Brief Title: Financial Incentives for Increasing Exercise
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped prior to recruitment due to logistical issues with the company in which it was going to be run.
Sponsor: Harvard University (Other)
Collaborators: Blue Cross Blue Shield (Other); Genzyme, a Sanofi Company (Industry); Partners HealthCare (Other)
Responsible Party: Michael I. Norton, Assistant professor of business administration, Harvard Business School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HBS-MN01
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2010-01

CONDITIONS: Sedentary Lifestyle; Obesity
Keywords: Sedentary lifestyle; physical exercise; behavioral economics; financial incentives; obesity
MeSH Terms: conditions — Sedentary Behavior; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (Experimental): 1) Control Group. Receives daily step goals via emails and has access to the study website to allow them to track their progress. Eligible for check-in incentives.
  Interventions: Behavioral: Financial incentives for increasing physical exercise
- Fixed (Experimental): Receives control intervention plus are incentivized to attain their daily step goals through daily lotteries:
  Each day, we will draw a two-digit number. If the first digit OR the second digit of this daily number matches the participant's lucky number, they win the small jackpot. If both digits match, they receive the large jackpot. Participants who meet their step goal for the day and who upload their data will be entered into the same lottery each day, where the small jackpot is $10 and the large jackpot is $100.
  Interventions: Behavioral: Financial incentives for increasing physical exercise
- Ascending (Experimental): Receives control intervention plus incentivized to attain daily step goals through lotteries:
  Each day, we will draw a two-digit number. If the first digit OR the second digit of this daily number matches the participant's lucky number, they win the small jackpot. If both digits match, they receive the large jackpot.
  Participants can increase their daily jackpots by meeting their step goals. Those who meet their goal for the first day of the week and who upload their data will be entered into a lottery where the small jackpot is $4 and the large jackpot is $40; if they successfully meet their step goal on the first day of the week, the jackpots for the second day increase to $6/$60, and so on such that if they reach their goals each day, the jackpots on day seven will reach $16/$160.
  Interventions: Behavioral: Financial incentives for increasing physical exercise
- Decreasing (Experimental): Receives control intervention plus incentivized to attain daily step goals through lotteries:
  Daily drawing procedure same as Ascending condition; structure of incentives is different: Participants can decrease their daily jackpots by failing to meet their step goals. Those who meet their goal for the first day of the week and who upload their data will be entered into a lottery where the small jackpot is $16 and the large jackpot is $160; if they successfully meet their step goal on the first day of the week, the jackpots will remain at $16/$160; if they do not meet their goal the jackpots will decrease to $14/$140, and so on such that if they fail to reach their goals each day, the jackpots on day seven will decrease to $4/$40.
  Interventions: Behavioral: Financial incentives for increasing physical exercise

INTERVENTIONS:
Behavioral: Financial incentives for increasing physical exercise — Throughout the 12-week intervention, participants will receive step goals. The step goals will increase by 250 steps per week, The intervention will last a total of 12 weeks. After each seven-day week, step goals will increase by an additional 250 steps - thus over the 12 weeks, participants will be asked to increase their daily step count by 3,000. Participants will receive financial incentives to attain these step goals; the incentive schemes differ according to intervention arm.

SUMMARY:
Participants will be employees of Genzyme who volunteer to participate in a study on motivating healthy behaviors, involving giving them goals for taking a certain number of steps per day, and increasing that number over time. Participants will wear pedometers and upload their data to a website that allows them to monitor their progress, and have the opportunity to win money based on meeting their step goals.

Interested employees will schedule a day and time to complete a health screening at a "Health Fair" at their place of employment, to ensure that they are healthy enough to participate; at this time participants will also complete the investigators baseline dependent measures, and receive a pedometer. After a one-week baseline period during which they wear the pedometer and the investigators establish their typical number of steps per day, eligible participants will then be assigned to one of four treatments - a "no incentive" control condition, and three conditions in which they are entered into different kinds of monetary lotteries if they have met their step goals for that day. Participants' initial goal will be based on their steps during the baseline period, and the goal will increase by 250 steps each week, for a total of 12 weeks. After these 3 months, the incentives portion of the experiment ends, but participants continue to wear their pedometers and upload their data for an additional 6 months. At 3 months, 6 months, and then at the study end at 9 months, participants again complete the investigators dependent measures at follow-up Health Fairs at their place of employment.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 28 or higher
* Pass the Par-Q
* answer "No" to all Par-Q questions
* at least 18 years of age
* has computer at home or work with compatible operating system (i.e. windows 2000, windows xp, windows vista, osX 10.3-10.5), internet access, and usb port

Exclusion Criteria:

* Anyone who does not meet all of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2013-04 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Physical activity | 12 weeks

SECONDARY OUTCOMES:
RAND 36-item Health Survey | 3mo, 6mo, 9mo
Health Stress questionnaire | 3mo, 6mo, 9mo
Emotional, Work, and Financial Attitudes questionnaire | 3mo, 6mo, 9mo
Weight loss | 3mo, 6mo, 9mo
Hemoglobin A1C | 6mo
Health behaviors questionnaire | 3mo, 6mo, 9mo
Word of mouth | 6mo, 9mo
Physical activity | 6mo, 9mo

CONTACTS AND LOCATIONS:
Overall Officials: Michael I. Norton, PhD, Principal Investigator — Harvard University
Locations (1):
- Genzyme, Cambridge, Massachusetts, United States